CLINICAL TRIAL: NCT02720250
Title: Effect of Omega-3 Fatty Acids Enriched Chicken Eggs Consumption on Microvascular Reactivity and Lipid Profile in Young Healthy Subjects
Brief Title: Omega-3 Fatty Acids Enriched Food and Microvascular Reactivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science, Faculty of Medicine Josip Juraj Strossmayer University of Osijek, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2158610714114
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Omega-3 Polyunsaturated Fatty Acids
Keywords: omega-3 fatty acids, microcirculation, laser Doppler flowmetry, lipid profile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Experimental): Intake of 3 omega-3 fatty acids enriched chicken eggs per day for three weeks.
  Interventions: Dietary Supplement: Omega-3 chicken eggs
- Regular (Experimental): Intake of 3 regular chicken eggs per day for three weeks.
  Interventions: Dietary Supplement: Regular chicken eggs

INTERVENTIONS:
Dietary Supplement: Omega-3 chicken eggs — Intake of 3 omega-3 fatty acids enriched chicken eggs per day for three weeks.
  Arms: Omega-3
Dietary Supplement: Regular chicken eggs — Intake of 3 regular chicken eggs per day for three weeks.
  Arms: Regular

SUMMARY:
Previous studies have shown that omega-3 fatty acid pills intake have beneficial effect on vascular health in overweight and/or hypertensive patients.

However, there is a lack of studies showing the effect of everyday consumption of omega-3 fatty acids enriched food (not pills) on lipid profile and microvascular reactivity in healthy population.

This study aimed to determine the effect of omega-3 enriched chicken eggs consumption on microvascular reactivity and lipid profile in young healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

- healthy volunteers

Exclusion Criteria:

* oral contraceptives
* drugs that could affect endothelium
* hypertension
* coronary artery disease
* diabetes
* hyperlipidaemia
* renal impairment
* cerebrovascular and peripheral artery disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
microvascular reactivity | Three weeks
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to vascular occlusion (post occlusive reactive hyperaemia - PORH) and in response to iontophoresis of acetylcholine (ACh) (endothelium dependent vasodilation).

SECONDARY OUTCOMES:
lipid profile | Three weeks
  Measurement of plasma cholesterol, HDL cholesterol, LDL cholesterol and triglycerides level.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Drenjancevic, MD, PhD, Principal Investigator — Faculty of Medicine, University of Osijek, Croatia
Locations (1):
- Faculty of Medicine Osijek, Laboratory for Clinical and Sport Physiology, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavka A, Cosic A, Jukic I, Jelakovic B, Lombard JH, Phillips SA, Seric V, Mihaljevic I, Drenjancevic I. The role of cyclo-oxygenase-1 in high-salt diet-induced microvascular dysfunction in humans. J Physiol. 2015 Dec 15;593(24):5313-24. doi: 10.1113/JP271631. Epub 2015 Dec 7. PMID 26498129